CLINICAL TRIAL: NCT04925713
Title: Phase 1 Trial of IFx-Hu2.0 to Evaluate Safety in Patients With Skin Cancer
Brief Title: IFx-Hu2.0 for the Treatment of Patients With Skin Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TuHURA Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC 2020-01
Expanded Access: NCT04853602 (Available)
Record Dates: First submitted 2021-06-02; First posted 2021-06-14 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2023-03

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Basal Cell Carcinoma
Keywords: cSCC; BCC; pAc/emm55; IFx-Hu2.0; Gene Therapy; Immunotherapy; Oncology; Immunology; plasmid DNA
MeSH Terms: conditions — Carcinoma, Basal Cell; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IFx-Hu2.0 (plasmid DNA) 0.1 mg/lesion (Experimental): One hundred (100) patients will receive 0.1 mg of IFx-Hu2.0 injected intratumorally in a single lesion at a single time point and be followed-up 28 days thereafter.
  Interventions: Biological: IFx-Hu2.0

INTERVENTIONS:
Biological: IFx-Hu2.0 — The investigational drug product IFx-Hu2.0 is composed of the drug substance pAc/emm55 (pDNA) complexed with the two excipients in vivo-jetPEI® (linear polyethylenimine), a transfection reagent, and dextrose, a pDNA/polyethylenimine complex stabilizer.
  Therapeutic Classification:
  * Immunomodulatory Agent
  Route of Administration:
  * Intralesional (i.e. injection of cutaneous, subcutaneous or lymph nodal lesions)
  Mechanism of Action:
  * Injection of IFx-Hu2.0 into the lesion facilitates the expression of the immunogenic Emm55 protein by the tumor cells.
  Physiological Effect:
  * Expression of the emm55 gene by the tumor cells triggers immune recognition of tumor-specific and -associated antigens which leads to innate and adaptive immune responses.
  Other Names: pAc/emm55

SUMMARY:
One hundred patients will receive IFx-Hu2.0 on an outpatient basis at a single time point in a single lesion. These patients will be assessed for any immediate adverse reactions and at Week 4 (Day 28+/-5 days) for any delayed adverse events..

DETAILED DESCRIPTION:
This is a multi-site, open-label, interventional, prospective, phase 1 trial to assess safety and tolerability of IFx-Hu2.0 in patients with basal cell carcinoma, squamous cell carcinoma, or cutaneous melanoma.

A total of approximately one hundred (100) male and/or female adult patients (greater than or equal to 18 years old), of any ethnicity and race, with at least one cutaneous melanoma, squamous cell carcinoma, or basal cell carcinoma lesion accessible for direct injection, who meet all inclusion and no exclusion criteria, will be eligible for enrollment and treatment with IFx-Hu2.0.

Enrollees will receive IFx-Hu2.0 as a single intralesional injection at a single time point. The target dose will be 100 μg of plasmid DNA per lesion injected at a final dose volume of 200 μL per lesion. The injected lesion will be completely excised at the follow-up visit four weeks later and will be biopsied for confirmation of diagnosis and for the establishment of a pathological response baseline peripheral blood will be collected from these patients prior to treatment administration and at the follow-up visit four weeks later. These samples will be used to perform complete blood counts (CBC) and clinical chemistry tests. A urine sample will be obtained for urinalysis for protein and blood at the same frequency. Blood samples will be drawn for immune response evaluation as well.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Ability to receive intralesional injections
4. Male or female, aged ≥ 18 years
5. Histologically confirmed cutaneous squamous cell carcinoma, or basal cell carcinoma with accessible lesions (based on archival tissue or new tissue biopsy for histological confirmation)
6. Life expectancy of at least 24 weeks at the time of screening
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
8. Must have measurable disease greater than 3 mm
9. At least one injectable lesion
10. Adequate organ function as defined below (Note: these screening laboratory tests must be obtained within two weeks prior to the baseline visit, Day 0):

    10.1. Hemoglobin (Hb) >10 g/dL 10.2. Absolute Neutrophil Count (ANC) >1,500 cells/mcL 10.3. Platelet Count (PLT) >75,000/mcL 10.4. Prothrombin Time (PT) or International Normalized Ratio (INR) ≤1.5 times the institutional ULN unless patient is receiving anticoagulant therapy as long as PT or INR is within therapeutic range of the intended use of anticoagulants.

    10.5. Activated Partial Thromboplastin Time (aPTT) ≤1.5 times the institutional ULN unless patient is receiving anticoagulant therapy as long as aPTT is within therapeutic range of the intended use of anticoagulants.

    10.6. Serum Creatinine (SCr) ≤1.5 times the institutional ULN 10.7. Total Bilirubin ≤1.5 times the institutional ULN 10.8. Aspartate Aminotransferase (AST) ≤3 times the institutional ULN 10.9. Alanine Aminotransferase (ALT) ≤3 times the institutional ULN 10.10. Lactate Dehydrogenase (LDH) ≤2 times the institutional ULN 10.11. Alkaline Phosphatase (ALP) ≤2.5 times the institutional ULN 10.12. Gamma GT (GGT) ≤2.5 times the institutional ULN
11. Lymphocyte count ≥500,000 cells/mL
12. For females of reproductive potential: must have a negative urine or serum pregnancy test result within 24 hours prior to receiving IFx-Hu2.0; must use highly effective contraception (e.g.,licensed hormonal or barrier methods) for at least one month prior to screening and agreement to use such a method during study participation and for an additional 26 weeks after the end of study treatment
13. For males of reproductive potential: use of barrier method or other methods to ensure effective contraception with partner

Exclusion Criteria:

1. Concurrent participation in any other clinical trial
2. Inability to consent for self
3. Lesions on scalp with bone erosions must not be selected as injection sites for IFx-Hu2.0
4. Life expectancy of fewer than 24 weeks at the time of screening
5. Prior systemic anti-cancer treatment within three weeks from start of treatment (Day 0)
6. Treatment with any investigational product within the three weeks preceding injection
7. Concurrent chemotherapy or biological therapy. Concurrent radiotherapy is allowed as long as it is not the same site as the injected lesion.
8. Current treatment with systemic immunosuppressive corticosteroid (greater than 10 mg of daily prednisone) doses or other immunosuppressants such as those needed for solid organ transplants. Medications needed to treat conditions such as reactive airway disease are not excluded.
9. Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 26 weeks after the last dose of trial treatment
10. Immunizations for encapsulated bacteria were not given for patients who have undergone a splenectomy
11. Serious underlying medical or psychiatric conditions, active infections requiring the use of antimicrobial drugs, or active bleeding that would make the subject unsuitable or unable to participate in the study
12. Active Human Immunodeficiency Virus (HIV)/Acquired Immunodeficiency Syndrome (AIDS) or Hepatitis B/C. Patients with treated HIV/AIDS or Hepatitis B/C with no evidence of active infection may be enrolled
13. History of organ allograft transplantation
14. Presence of any uncontrolled and significant medical or psychiatric condition which would interfere with trial safety assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Moore Clinical Research, Brandon, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion: Biological: IFx-Hu2.0 The investigational drug product IFx-Hu2.0 is composed of the drug substance pAc/emm55 (pDNA) complexed with the two excipients in vivo-jetPEI® (linear polyethylenimine), a transfection reagent, and dextrose, a pDNA/polyethylenimine complex stabilizer.
  Therapeutic Classification:
  Immunomodulatory Agent
  Route of Administration:
  Intralesional (i.e. injection of cutaneous, subcutaneous or lymph nodal lesions)
  Mechanism of Action:
  Injection of IFx-Hu2.0 into the lesion facilitates the expression of the immunogenic Emm55 protein by the tumor cells.
  Physiological Effect:
  Expression of the emm55 gene by the tumor cells triggers immune recognition of tumor-specific and -associated antigens which leads to innate and adaptive immune responses.
  Other Name: pAc/emm55
Period: Overall Study
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Cutaneous Squamous Cell Carcinoma [Count of Participants; unit: Participants] | 2
Basal Cell Carcinoma [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Adverse Events
Description: Rate of Adverse Events reported per Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Time Frame: 28 days post injection
Measure: Count of Participants; unit: Participants
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion
Number analyzed (Participants) | 5
Participants
  Serious Adverse Events (SAEs) | 0
  Dose Limiting Toxicity (DLT) | 0
  Participants Analyzed | 5

2. Primary Outcome: Number of Patients Who Completed the Trial [Time Frame: 28 Days Post Injection]
Description: Number of Patients who completed the trial per protocol without major deviations.
Time Frame: 28 days post injection
Measure: Count of Participants; unit: Participants
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion
Number analyzed (Participants) | 5
Participants
  Number of Patients who completed the trial | 5
  Number of Patients who did not completed the trial | 0

ADVERSE EVENTS:
Time Frame: Day 0 to 28 days ± 7 business days from the last dose administered.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion: 0.1 mg of IFx-Hu2.0 injected intratumorally in a single lesion at a single time point and with a follow up visit 28 days thereafter.
Arm/Group | IFx-Hu2.0 (Plasmid DNA) 0.1 mg/Lesion
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT04925713/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/13/NCT04925713/SAP_001.pdf